CLINICAL TRIAL: NCT02858830
Title: Genetic and Metabolic Basis of Familial Partial Lipodystrophy
Brief Title: Familial Partial Lipodystrophy Study
Acronym: FPL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Vinaya Simha, M.B.B.S., M.D., PI, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-009144
Record Dates: First submitted 2016-05-19; First posted 2016-08-08 (Estimated); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Lipodystrophy, Familial Partial
Keywords: FPL; adipose tissue; diabetes; dyslipidemia; metabolic; hyperinsulinemia
MeSH Terms: conditions — Lipodystrophy, Familial Partial; Diabetes Mellitus; Dyslipidemias; Hyperinsulinism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: Healthy Subject (Other): Healthy Subject (Control) will undergo assessments before and after ingesting a high fat mixed meal.
  Interventions: Other: High fat mixed meal
- Group 2: FPL Subject (Other): FPL Subject will undergo assessments before and after ingesting a high fat mixed meal.
  Interventions: Other: High fat mixed meal

INTERVENTIONS:
Other: High fat mixed meal

SUMMARY:
Studying patients with rare adipose tissue disorders may help the investigators to better understand the pathophysiology of diabetes and dyslipidemia in relation to adiposity, and thus have an enormous impact on public health.

DETAILED DESCRIPTION:
A systematic study of body fat distribution is necessary to better define the phenotypic spectrum of FPL, and to better recognize FPL in patients with Metabolic Syndrome. Similarly, genetic studies in these patients will not only help better characterize the genotype-phenotype relationship, but is also likely to help identify other genes involved in regulation of lipid homeostasis, as some patients may not have any of the known mutations.

The Investigators will systematically study mitochondrial protein quality and function under fasting and fed state in relation to intramyocellular and circulating plasma lipid levels, and compare with age, sex and BMI-matched individuals. The Investigators will also study the rate of de-novo protein synthesis to determine if hyperinsulinemia affects both muscle protein anabolism and catabolism.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of lipodystrophy (decreased subcutaneous fat)
2. Family history of lipodystrophy
3. Normal control subject

Exclusion Criteria:

1. Inability to provide informed consent
2. Hemoglobin < 10g%

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-08; Primary Completion 2017-04-14 (Actual); Study Completion 2017-04-14 (Actual)

PRIMARY OUTCOMES:
Upper body muscle strength measured by chest press dynamometry | Before consumption of a high fat mixed meal
Change in fractional mitochondrial protein synthesis rates | Before and after consumption of a high fat mixed meal (approximately 4 hours after the meal)
Lower body muscle strength measured by knee extension | Before consumption of a high fat mixed meal

CONTACTS AND LOCATIONS:
Overall Officials: Vinaya Simha, MBBS, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials